CLINICAL TRIAL: NCT03114787
Title: Does Respiratory Physiotherapy Allow for Earlier Withdrawal of Mechanical Ventilation in Respiratory Resuscitation Service? Randomized Controlled Trial
Brief Title: Does Respiratory Physiotherapy Allow for Earlier Withdrawal of Mechanical Ventilation in Respiratory Resuscitation Service?
Acronym: KISEVEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient recruiting was stopped after 17 inclusions because of a reorganization of Intensive Care Units at the recruiting center.
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0014
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Physiotherapy; Resuscitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient receiving respiratory physiotherapy (Other)
  Interventions: Other: Study on patients with respiratory resuscitation
- Patient not receiving respiratory physiotherapy (Other)
  Interventions: Other: Study on patients with respiratory resuscitation

INTERVENTIONS:
Other: Study on patients with respiratory resuscitation — Patient intubated with mechanical ventilation in VS-AI mode, whose weaning is difficult

SUMMARY:
Respiratory physiotherapy is not routinely prescribed in the resuscitation department and few studies deal with this subject, especially in respiratory resuscitation

ELIGIBILITY:
Inclusion Criteria:

* Patient intubated with mechanical ventilation in VS-AI mode, whose weaning is difficult
* Major Patient over 18 years of age
* Patient affiliated to social security

Exclusion Criteria:

* Sedate
* With restrictive or tracheotomized syndrome
* With rib fractures
* Not able to benefit from physiotherapy within 3 hours after the start of the weaning protocol
* Refusal of patient or family
* Physiotherapy contraindications
* Patient under tutorship or curatorship
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Time between initiation of weaning protocol and extubation. | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France